CLINICAL TRIAL: NCT04704310
Title: Enhancing Exercise Training for Adults With COPD: The Roles of Peers and Functional Tasks
Brief Title: Enhancing Exercise Training for Adults With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Fondation Québécoise en Santé Respiratoire (Unknown)
Responsible Party: Principal Investigator, Shane Norman Sweet, Associate Professor, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 250956
Record Dates: First submitted 2020-12-22; First posted 2021-01-11 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: exercise; peer support; behavior change
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Intervention Model Description: A convenience sample of adults living with COPD (N=4-6) will be recruited to participate an 8- week online exercise intervention.The objective is to conduct a proof-of-concept online exercise intervention for individuals living with COPD, using functional tasks, and incorporating peer support.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Individuals acting as own control. Looking at changes pre and post intervention
  Interventions: Behavioral: Enhancing exercise training for adults with COPD: The roles of peers and functional tasks

INTERVENTIONS:
Behavioral: Enhancing exercise training for adults with COPD: The roles of peers and functional tasks — A proof-of-concept online 8-week exercise training program for adults with COPD that incorporates both a peer mentorship and a functional tasks component.

SUMMARY:
This study aims to find a new way to get individuals living with COPD to become and stay active during and after an exercise intervention. In this study, individuals living with COPD will participate in an online exercise intervention. The exercises included in this intervention are based in individuals' activities of daily living. Additionally, during this intervention, individuals with COPD will participate in peer support sessions and will be taught and encouraged to discuss eight behaviour change techniques that have been shown to help support increased participation in physical activity and/or exercise. The goal of this study is to test out this new protocol and determine if it is feasible to recreate on a larger scale and if it is acceptable for the COPD community.

ELIGIBILITY:
Inclusion Criteria: Individuals must be at least 18 years of age, have no diagnosed cognitive impairment, have a COPD diagnosis (any stage), be medically able to participate in exercise (confirmed by healthcare professional in the past 2 years), have access to a computer with a camera and internet, and speak English or French.

Exclusion Criteria: less than 18 years of age, diagnosed with a cognitive impairment, not diagnosed with COPD by a medical professional, unable to participate in exercise or unconfirmed in the past 2 years from a medical professional, no access to a computer and internet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Participant Adherence | 8 weeks
  Intervention adherence will be measured be taking attendance for each session (2 x 8 weeks = 16 sessions). Intervention feasibility as an indicator of success will be an overall program adherence rate of 70% (approximately 11 sessions attended by all participants, respectively)
Participant Engagement | 8 weeks
  Participant engagement will be measured by counting the number of unique topics brought up by each participant. The indicator of success will be that each participant initiates 1 topic of conversation in 70% of session (initiates 11 conversations during program)
Goal Participation | 8 weeks
  Participant goal participation will be measured by improvement in initial goals set at the beginning of the study using the Canadian Occupation Performance Measures (COPM). Success will be determined by calculating individuals change score on their satisfaction with their performance in their target areas. A change score of 2 on an item is said to represent significant change (Law et al., 2000). A change score of at least 2 on 50% of items (dependent on personal goals) for 70% of participants will be the indicator of success.

SECONDARY OUTCOMES:
Timed "Up & Go" test | Baseline, immediately after intervention (9 weeks after baseline)
  This test measures the time it takes an individual to stand from a standard chair (approximately 46cm), walk 3 metres, walk back, and return to sit on the chair (Podsiadlo & Richardson, 1991). The participant is timed from when the leave the seat to when they are seated again. A time of >30 seconds is the cut-off for safe unsupervised participation (Podsiadlo & Richardson, 1991). Anyone who gets a time >30seconds will be informed that they cannot participate.
1-minute sit-to-stand test | Baseline, immediately after intervention (9 weeks after baseline)
  This test is a measure of exercise capacity that has been validated with individuals living with COPD (Puhan et al., 2013). Individuals sit on a standard chair without arm rests, keep their legs apart with about 90 degrees knee flexion and aligned with their hips, and are asked to hold their hands stationary on their hips.For the duration of 1 minute, participants are asked to do as many repetitions as possible of the sit to stand, without using arms for support. The number of repetitions is recorded.
Handgrip Test | Baseline, immediately after intervention (9 weeks after baseline)
  A Hand Dynamometer was be used to measure handgrip strength. Individuals sit with their shoulders adducted, elbows flexed to 90 ̊ and forearms in a neutral position (Puhan et al., 2013). They are then asked to squeeze the handle as much as possible and read to the nearest kilogram where the needle stopped, which is recorded. The best of six measurements is used as an indication of upper body strength.
Six-minute walk test | Baseline, immediately after intervention (9 weeks after baseline)
  To perform the six-minute walk test, participants walk along a track (or hallway) that is a minimum of 25 meters long (marked at each meter). Participants are instructed to walk at a comfortable pace for six minutes. Participants' dyspnea score will be measured using the modified Borg scale (Kendrick et al., 2000). A lower score, or covering less distance during the six minutes, is indicative of worse physical endurance and function (Sciurba et al., 2003). The distance walked by each participant during the six minutes is recorded after each test.
  If participants do not have a hallway that is 25 meters long, participants are asked to run/walk as far as possible in 6 minutes, tracking the number of steps they take or distance travelled with a free application on their phone. Take pulse immediately after completing the exercise for 1 minute (determine bpm).
3-minute step test | Baseline, immediately after intervention (9 weeks after baseline)
  An alternative for the 6-minute walk/run test that can be completed indoors. Participants' will step up onto a single step and then back down repeatedly for 3 minutes. To determine beats per minute (BPM), take pulse immediately after completing the exercise for 1 minute. Participants' dyspnea score will be measured using the modified Borg scale (Kendrick et al., 2000). Number of steps is also recorded (Beaumont et al., 2019). Results are relative to the individual but provides a good indication of aerobic fitness and can be used to track progress.
Borg Scale - Dyspnea | Baseline, immediately after intervention (9 weeks after baseline)
  On a scale from 0-10, participants' indicate their breathlessness level. 0- No breathlessness at all to 10- Maximal breathlessness
Motivation for Exercise Questionnaire | Baseline, immediately after intervention (9 weeks after baseline)
  This questionnaire was used to measure participants' reasons is for why they are, or would like to be, active on a regular basis. The rating scale is 1-7, 1 being not true at all, and 7 being very true
Godin Leisure Time Physical Activity Questionnaire | Baseline, immediately after intervention (9 weeks after baseline)
  Self-reported physical activity levels measured in length of bouts over the previous 7 days to determine physical activity frequency.
The Psychological Need Satisfaction in Exercise scale | Baseline, immediately after intervention (9 weeks after baseline)
  This 1-6 scale represents different feelings people have when they exercise. 1-true to how they typically feel when exercising, and 6-false to how they typically feel when exercising.
The Satisfaction with Life Questionnaire | Baseline, immediately after intervention (9 weeks after baseline)
  This 5 item questionnaire was used to measure participants' level of life satisfaction. The higher the score, the higher the sense of life satisfaction. A score from 5-9 indicated extremely dissatisfied, 10-14 is dissatisfied, 15-19 indicated slightly below average life satisfaction. 20-24 is the average score, 25-29 is a high score indicative of higher life satisfaction and a score between 30-35 is a very high score and represent very high life satisfaction.

OTHER OUTCOMES:
COPD Assessment Test (CAT) | Baseline, immediately after intervention (9 weeks after baseline)
  This questionnaire was used to measure the impact COPD is having on well being and daily life. The CAT is an eight-item semantic differential scale from 0 to 5, where 0 is no impact and 5 is extremely impactful. Items include: I never cough| I cough all the time, I have no phlegm (mucus) in my chest at all | My chest is completely full of phlegm (mucus), My chest does not feel tight at all | My chest feels very tight, When I walk up a hill or one flight of stairs, I am not breathless | When I walk up a hill or one flight of stairs, I am very breathless, I am not limited doing any activities at home| I am very limited doing activities at home, I am confident leaving my home despite my lung condition| I am not at all confident leaving my home because of my lung condition, I sleep soundly | I don't sleep soundly because of my lung condition, I have lots of energy I have no energy at all. Participants' scores were totaled and a score of ≥ 10 indicated higher than normal burden of disease.
Medical Research Council Questionnaire on Breathlessness | Baseline, immediately after intervention (9 weeks after baseline)
  This questionnaire was used to measure participants' breathlessness burden using a single item scale from 0 to 4, where a score of 0-1 indicated mild breathlessness and 2-4 indicated increased breathlessness.

CONTACTS AND LOCATIONS:
Overall Officials: Shane N Sweet, Ph.D, Principal Investigator — McGill University
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No